CLINICAL TRIAL: NCT03534817
Title: Early Versus Standard Access Cardiac Rehabilitation to Counter Ventricular Remodeling Post-MI (EVADE): a Pilot-Feasibility Study.
Brief Title: Early Versus Standard Access Cardiac Rehabilitation to Counter Ventricular Remodeling Post-MI (EVADE)
Acronym: EVADE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: University of Saskatchewan (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Saskatchewan Health Research Foundation (Other); Royal University Hospital Foundation (Other); University of Alberta (Other)
Responsible Party: Principal Investigator, Corey Tomczak, Assistant Professor, College of Kinesiology, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: USaskatchewan-EVADE
Record Dates: First submitted 2018-01-16; First posted 2018-05-23 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Myocardial Infarction
Keywords: Cardiac Rehabilitation; Early Access Cardiac Rehabilitation; Cardiac Rehabilitation Adherence; Myocardial Infarction; Ventricular Remodeling
MeSH Terms: conditions — Myocardial Infarction; Ventricular Remodeling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Access CR (Experimental): Participants begin cardiac rehabilitation (CR) after 1-week following discharge post-MI.
  Interventions: Behavioral: Early Access CR
- Standard Access CR (No Intervention): Participants begin CR after 7-weeks following discharge post-MI, similar to the average Canadian wait time.

INTERVENTIONS:
Behavioral: Early Access CR — Participants in the Early Access CR group will begin CR within 1-week post-hospital discharge following their MI, as opposed to Standard Access CR group which begins 7-weeks post-hospital discharge, and the Canadian average (10-14 weeks post-hospital discharge). No further intervention or differentiation between groups is applied; the actual CR program is standardized between groups, and follows the guidelines regularly practiced by the institution.
  Arms: Early Access CR

SUMMARY:
BACKGROUND: Cardiac rehabilitation (CR) is an outpatient chronic disease management program delivering secondary prevention, which is proven to reduce morbidity and mortality. The Canadian Cardiovascular Society Access to Care working group recommends patients access CR "preferably" within 2-7 days following percutaneous intervention for myocardial infarction (MI), but that 30-60 days is "acceptable". Despite these benchmarks, in practice patients access CR up to 90 days post-treatment in Canada. This is disconcerting given the detrimental impacts of delayed access to CR. These include ventricular remodeling (i.e., ventricular enlargement and reduced pump function), lower CR use, less post-CR exercise, among others. Accordingly, EVADE will be the first randomized controlled trial (RCT) to test the effects of early access CR (1-week post-discharge to first CR visit) compared to standard access CR (7-weeks post-discharge to first CR visit) in ameliorating these concerns.

AIMS & HYPOTHESIS: The primary aim is to compare ventricular remodeling as defined by the change in end-systolic volume at 1-year in participants randomized to early versus standard access CR. The secondary aims are: (1) to compare post-CR exercise adherence by accelerometry, exercise capacity by 6-minute walk test distance, and health-related quality of life (HRQL) at 1-year in participants randomized to early versus standard access CR; (2) to compare CR program session attendance in participants randomized to early versus standard access CR; and (3) to assess biomarkers of ventricular remodeling in participants randomized to early versus standard access CR.

The final aims are to explore more immediate health benefits associated with early versus standard access CR. Accordingly, at 6 months following hospital discharge the investigators will measure end-systolic volume, exercise adherence, exercise capacity, biomarkers of ventricular remodeling, and HRQL. The investigators will also explore hospitalization for any cause of death at 1 year in order to inform future research.

The overall hypothesis is that early access CR will be associated with less ventricular remodeling, increased CR attendance and post-CR exercise adherence, increased exercise capacity, and greater HRQL.

DESIGN: EVADE will be a two-centre, 2 parallel-arm, single-blinded RCT. Participants will be recruited through coronary care units following treatment for MI from the Royal University Hospital in Saskatoon, Saskatchewan and the University of Alberta Hospital in Edmonton. The University of Alberta Research Electronic Data Capture (REDCap) online database will randomize (1:1) participants (allocation concealed). A total of 60 participants will be enrolled: 30 participants will each be allocated to early access and standard access CR.

IMPACT: In the first prospective multicentre trial of its kind, EVADE will test an innovative post-MI rehabilitation strategy that has the potential to demonstrate the superior benefits of early access CR for attenuating ventricular remodeling, and increasing CR attendance, post-CR exercise adherence, exercise capacity, and HRQL. The results from EVADE would encourage the Canadian CR community to consider early access CR to further enhance readily available and existing CR programs. The knowledge gained from EVADE will inform clinical decision-making practices, influence future CR guidelines and policy, and will contribute to the ongoing goal of improving efficiency and effectiveness of the Canadian health care system.

ELIGIBILITY:
Inclusion Criteria:

* have a cardiologist-diagnosed non ST-segment elevation MI (NSTEMI) or ST-segment elevation MI (STEMI) identified as low risk based on the Global Registry for Acute Coronary Events (GRACE) risk score;
* have angiographic evidence of revascularization of the infarct-related artery that is defined as ≥80% patency;
* have an ejection fraction ≥35% (to exclude patients needing a cardioverter defibrillator) and <50% (consistent with impaired heart pump function);
* reside within 100 km (1 hour travel time) of Saskatoon/Edmonton city limits;
* have been approved to attend CR by their attending physician.

Exclusion Criteria:

* have been hospitalized for a previous MI
* have a condition that precludes walk testing;
* have a contra-indication for cardiac MRI (i.e., pacemaker, pregnancy);
* index hospitalization >10 days;
* undergo coronary artery bypass grafting;
* does not undergo coronary angiography.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in ventricular remodeling from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | A repeated measures approach will be taken for the primary outcome: before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI.
  End-diastolic volume (in milliliters) will be the primary marker of ventricular remodeling, and will be measured using clinical-grade cardiac magnetic resonance imaging (MRI).

SECONDARY OUTCOMES:
Change in end-systolic volume (in milliliters) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  End-systolic volume will indicate change in ventricular systolic function, which in turn indicates functional ventricular remodeling. End-systolic volume will be measured using clinical-grade cardiac magnetic resonance imaging (MRI).
Change in stroke volume (in milliliters) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  Stroke volume will indicate change in ventricular function, which in turn indicates functional ventricular remodeling. Stroke volume will be measured using clinical-grade cardiac magnetic resonance imaging (MRI).
Change in ejection fraction (percentage) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  Ejection fraction will indicate change in ventricular function, which in turn indicates functional ventricular remodeling. Ejection fraction will be measured using clinical-grade cardiac magnetic resonance imaging (MRI).
Change in MI-related cardiac damage from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  MI-related cardiac damage will be measured using clinical-grade cardiac magnetic resonance imaging (MRI).
Change in metalloproteinase-9 (MMP-9) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  MMP-9 levels (nanogram/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
Change in high-sensitivity C-reactive protein (hsCRP) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  hsCRP levels (milligram/liter) will be analysed from blood samples taken by a registered phlebotomist.
Change in brain-type natriuretic peptide (BNP) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  BNP levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
Change in soluble receptor for advanced glycation end-products (sRAGE) from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  sRAGE levels (picograms/milliliter) will be analysed from blood samples taken by a registered phlebotomist.
Change in exercise capacity from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  Participants will complete a 6-minute walk test; participants will walk for 6 minutes and will be encouraged to walk as fast as possible without running. The distance covered will be their score.
Change in perceived health-related quality of life from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI.
  The Short Form Health Survey (SF-36) evaluates and scores a participant's perceived quality of life with a numerical score on a scale. The overall score (range 0-100, mean) is an average of the subscales, which include the physical function score (range 0-100, mean of scores), quality of life limitations due to physical health (range 0-100, mean of scores), quality of life limitations due to emotional problems (range 0-100, mean of scores), energy levels score (range 0-100, mean of scores), emotional well-being (range 0-100, mean of scores), social functioning (range 0-100, mean of scores), pain (range 0-100, mean of scores), and general health (range 0-100, mean of scores). For the overall scale and the subscales, a higher value represents higher perceived health-related quality of life and a better outcome.
Change in heart-related anxiety from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI.
  The Heart-Related Anxiety questionnaire evaluates and scores a participant's perceived anxiety related to their heart condition with a numerical score on a scale. The scale has 18-items scoring 0-4, and the measure's total score is the sum of scores (range 0-72) with a lower score representing less anxiety and a better outcome.
Change in hospital-related anxiety and depression from in-hospital following MI to 6-months (immediate change) and 12-months post-MI (long-term change). | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI.
  The Hospital Anxiety and Depression Scale (HADS) evaluates and scores a participant's perceived anxiety and depression following hospitalization with a numerical score on a scale. The questionnaire has 14-items total, 7 anxiety and 7 depression related questions, each scoring 0-3. The questionnaire has two subscales; anxiety (range 0-21) and depression (0-21). The item scores are summed to give the subscale score, with a lower value representing less anxiety or less depression and better outcomes.
Exercise history | On the first visit to CR.
  The Godin Leisure Time Exercise Questionnaire (modified) scores a participant's recreational physical activity levels outside of employment within the past 4 weeks. This questionnaire will capture and account for physical activity performed prior to commencing CR. This questionnaire is not a scale as it does not have a maximum value, thus the range is not provided. It provides a score based by summing the number of bouts of light, moderate, and heavy physical activity, increasing the relative contribution of exercise intensity by adding a multiplier to the number of exercise bouts depending upon the intensity (i.e., multiply by 9 for heavy, by 5 for moderate, and by 3 for light activity). E.g., With 3 heavy exercise sessions, 6 moderate sessions, and 14 light sessions, the total leisure activity score = (9 × 3) + (5 × 6) + (3 × 14) = 27 + 30 + 42 = 99. A higher score represents a greater physical activity volume and a better outcome.
Change in post-CR exercise adherence (exercise duration in minutes) from the end of the 3 month CR program, to 6-months (immediate change), 9-months (immediate change), and 12-months post-MI (long-term change). | Before the end of 3 month CR program (within the last two weeks of their program); at 6 months post-MI; at 9-months post-MI; at 12 months post-MI.
  Tri-axial accelerometers will be worn for 7 consecutive days, 24 hours a day. The average daily minutes of moderate-to-vigorous physical activity will be recorded and calculated.
Change in post-CR exercise adherence (daily steps) from the end of the 3 month CR program, to 6-months (immediate change), 9-months (immediate change), and 12-months post-MI (long-term change). | Before the end of 3 month CR program (within the last two weeks of their program); at 6 months post-MI; at 9-months post-MI; at 12 months post-MI.
  Tri-axial accelerometers will be worn for 7 consecutive days, 24 hours a day. The average daily minutes of moderate-to-vigorous physical activity will be recorded and calculated.
CR Attendance | At the end of 3 month CR program.
  Participants attendance will be recorded as number of session per week.
CR Adherence | At the end of 3 month CR program.
  Participants will keep a log of their CR exercise type, duration, and intensity which will be given to investigators at the end of the CR program.
Hospitalization | 12-months post-MI.
  During the final data collection visit, the participant will report all unanticipated hospital and emergency department visits during the last year since their MI. Study investigators will also do a search in the health region of hospitalization and emergency visits.
Death | 12-months post-MI.
  If the participant has deceased prior to the end of the trial (i.e., 12-months post MI), this will be recorded.

OTHER OUTCOMES:
Infarction Type | Before hospital discharge
  The type of infarction (STEMI vs. NSTEMI) will be used to stratify patients between the two treatment arms.
Medications | Before hospital discharge and 12 months post-MI
  Medications will be recorded for participant characteristic data.
Medical History | Before hospital discharge and 12-months post-MI
  Medical history will be recorded for participant characteristic data.
Height in meters | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  Height will be gathered as participant characteristic data in a repeated measures approach.
Weight in kilograms | Before hospital discharge following MI; at 6 months post-MI; at 12 months post-MI
  Weight will be gathered as participant characteristic data in a repeated measures approach.

CONTACTS AND LOCATIONS:
Overall Officials: David (Ian) Paterson, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No